CLINICAL TRIAL: NCT02033460
Title: Manual Therapy vs Manual Therapy and Exercise vs Manual Therapy and Exercise and Education in Patients With Chronic Neck Pain
Brief Title: Manual Therapy Versus Manual Therapy and Exercise and Education in Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Josue Fernandez Carnero (Other)
Collaborators: Universidad Autonoma de Madrid (Other)
Responsible Party: Sponsor-Investigator, Josue Fernandez Carnero, Associate Professor, Universidad Rey Juan Carlos
Organization: Universidad Rey Juan Carlos (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PI-551
Record Dates: First submitted 2014-01-09; First posted 2014-01-10 (Estimated); Last update posted 2014-01-13 (Estimated); Status verified 2014-01

CONDITIONS: Neck Pains; Posterior Cervical Pains; Posterior Neck Pain; Cervicalgia
Keywords: Manual therapy; Exercise; Education
MeSH Terms: conditions — Neck Pain; Motor Activity | interventions — Musculoskeletal Manipulations; Educational Status; Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Manual therapy, education and Exercise (Experimental): The protocol for this group is identical to the previous group with the sole difference that is added an exercise protocol :
  In the fifth session we explained the patients to perform :
  * Five sets of isometric contraction of the deep neck flexors for 8-10 seconds.
  * Five sets of isometric contraction of the neck extensors for 6-8 seconds
  * Neural self-mobilization and stretching held for 10 - 12 seconds for the levator scapulae and the trapezius muscle.
  In the sixth session the patient repeat all the exercises from the previous session and also with the help of a theraband made :
  • Isotonic contraction of the head, performing 3-4 sets of 8-10 repetitions.
  Interventions: Other: Manual Therapy and Education; Other: Manual Therapy
- Manual Therapy and Education (Active Comparator): The protocol used for therapeutic education consisted of two approaches:
  Manual therapy will consist on Traction oscillatory,craniocervical region, Mobilization of upper cervical region in flexion, Side glide roll, Mobilization upper cervical anteroposterior with Wedge, Sliding lateral techniques and High-velocity technique in dorsal region. And Education of the physiology of pain and Education about cognitive behavioral perspective.
  Interventions: Other: Manual Therapy; Other: Manual therapy, Education and Exercise
- Manual Therapy (Active Comparator): Manual therapy will consist on Traction oscillatory, Mobilization of upper cervical region in flexion, Side glide roll, Mobilization upper cervical anteroposterior with Wedge, Sliding lateral C1- C2 ( 2 minutes) , C2 -C3, and C5 -C6 and High-velocity technique in dorsal region.
  Interventions: Other: Manual Therapy and Education; Other: Manual therapy, Education and Exercise

INTERVENTIONS:
Other: Manual Therapy and Education — Manual therapy will consist on Traction oscillatory,craniocervical region, Mobilization of upper cervical region in flexion, Side glide roll, Mobilization upper cervical anteroposterior with Wedge, Sliding lateral techniques and High-velocity technique in dorsal region. And Education of the physiology of pain and Education about cognitive behavioral perspective will add to manual therapy treatment.
  Arms: Manual Therapy; Manual therapy, education and Exercise
Other: Manual Therapy — Manual therapy will consist on Traction oscillatory, Maintained traction in the craniocervical region, Mobilization of upper cervical region in flexion, Side glide roll, Mobilization upper cervical anteroposterior with Wedge, Sliding lateral C1- C2 ( 2 minutes) , C2 -C3, and C5 -C6 and High-velocity technique in dorsal region.
  Arms: Manual Therapy and Education; Manual therapy, education and Exercise
Other: Manual therapy, Education and Exercise — Manual therapy will consist on Traction oscillatory,craniocervical region, Mobilization of upper cervical region in flexion, Side glide roll, Mobilization upper cervical anteroposterior with Wedge, Sliding lateral techniques and High-velocity technique in dorsal region. And Education of the physiology of pain and Education about cognitive behavioral perspective and Craniocervical exercise will add to this arm.
  Arms: Manual Therapy; Manual Therapy and Education

SUMMARY:
The purpose of this study is to know which combination of treatments are the most effective in patients with non-specific neck pain. Study design: This is a single-blind randomized controlled trial. (outcomes assessor). Study population: Men and women aged 18 to 60 years old with neck pain for at least 12 weeks. Interventions: 3 groups will be treated for a period of 4 weeks (8 sessions total; 2 per week).

DETAILED DESCRIPTION:
Nonspecific chronic neck pain has a high prevalence and is very common in clinical practice.

Manual therapy (MT) studies of techniques like mobilization, manipulation, and therapeutic exercise, has been demonstrated effectiveness for the treatment of pain and disability in the neck. These investigations have thought of this treatments as individual interventions. Thus, multimodal ways of treatment to improve patients with nonspecific chronic neck pain are necessary.

The aim of this study is to evaluate the effectiveness of a multimodal treatment protocol compared to a unimodal treatment protocol in the medium-term, on patients with chronic non-specific neck pain.

Subjects are randomly allocated into three groups: MT group; MT+Educational therapy (ET) group; and MT+ET+Exercise group. Each subject receive a 4 weeks period treatment (8 sessions). Outcome measures include physical, somatosensory, and psychosocial characteristics; which are measure at 0, 4, 8, 16 weeks by a blinded assessor.

ELIGIBILITY:
Inclusion Criteria:

* The subjects for the study were selected if they fulfilled the following inclusion criteria: Aged between 18 to 60 years old, head and/or neck pain for at least 12 weeks and having the willing to undergo the treatment.

Exclusion Criteria:

* if they had appearance of "red flags", rheumatologic diseases or any type of cancer, cervical surgery in the past, whiplash trauma and undergoing any type of treatment like physical therapy, manual therapy, osteopathy, chiropraxis, acupuncture during the last three months. All patients recruited for the study complained of pain localized in the neck and/or head region. Initial screening was accomplished by telephone and eligible persons attended a evaluation appointment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-01; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
visual analogue scale | pre-treatment, 4, 8, 16 weeks
  This scale comprises of a 100-mm horizontal line with pain descriptors marked "no pain" at left side and "the worst pain imagine" at the right side, and is used to measure the pain intensity. It was recorded at the beginning of the physical assessment and the patient was asked what their pain intensity was at the time by marking the VAS with a perpendicular line. This is a valid method to measure the pain level37 and psychometric properties of the VAS have been reported widely. The minimal important difference of the VAS is based on detecting an 8.6 mm (based in previous study for a score < 40mm with a pain onset more than 12 weeks) of difference immediately after treatment.
Pressure Pain threshold | pre-treatment, 4, 8, 16 weeks
  Pressure pain threshold (PPT) is defined as the amount of pressure where the sense of pressure first changes to pain. A digital algometer (FDX 25, Wagner Instruments, CT, USA), will be used. Pressure pain threshold was assessed over right side of masseter 1 and 2, the temporalis muscle 1 and 2, suboccipital muscle, spinous process of C2, vertebral joint process of C5 y C6, upper trapezius muscle (midway between C7 and acromion), epicondyle, scaphoid bone and tibialis anterior muscle (upper one-third of the muscle belly) by an assessor blinded to the subject's condition.
Cervical Range of Motion | pre-treatment, 4, 8, 16 weeks
  Cervical spine mobility was measured with Cervical Range of Motion (CROM) device (Performance Attainment Associates, MN). The CROM is an instrument that assesses the active range of motion of the cervical segment. It´s a reliable method of measuring, providing a range of intra-meter reliability from 0.7 to 0.9 and a range of inter-meter reliability from 0.8 to 0.87. The patients were measured while sitting with the back against a chair. The goniometer placed over his head, is asked to perform analytical neck movements (flexion, extension, right lateral flexion, left lateral flexion, right rotation and left rotation).
Neck disability index | pre-treatment, 4, 8, 16 weeks
  It is a well-validated 10-item questionnaire. The Neck Disability Index (NDI) has sufficient support in the literature, to be the most commonly used to report neck pain. It was used a spanish validation of the index. Scores of <4 indicate no disability, 5-14 mild disability, 15-25 moderate disability, 25-34 severe disability and >35 complete disability

SECONDARY OUTCOMES:
Kinesiophobia | Pre-treatment, 4, 8, 16 weeks
  The Tampa Scale for Kinesiophobia, developed by Miller was used to assess fear of movement and injury. We used a 11-items version.
Catastrophizing | Pre-treatment, 4, 8, 16 weeks
  To evaluate the subject's propensity to catastrophize about pain we used the Spanish version of Pain Catastrophizing Scale (PCS). This scale is a 13-item questionnaire designed to measure the three components of catastrophizing: rumination, magnification and helplessness, resulting this evaluation in a unique score.
Fear Avoidance Belief Questionnaire (FABQ) | Pre-treatment, 4, 8, 16 weeks
  The FABQ assesses patient beliefs with regard to the effect of physical activity and work on their pain. It consists of 16 items and patients rate their agreement with each statement on a 7- point Likert scale (0 = completely disagree, 6 = completely agree).

CONTACTS AND LOCATIONS:
Overall Officials: Josue Fernandez-Carnero, PhD, Study Director — Universidad Rey Juan Carlos

REFERENCES:
- [Derived] Beltran-Alacreu H, Lopez-de-Uralde-Villanueva I, Fernandez-Carnero J, La Touche R. Manual Therapy, Therapeutic Patient Education, and Therapeutic Exercise, an Effective Multimodal Treatment of Nonspecific Chronic Neck Pain: A Randomized Controlled Trial. Am J Phys Med Rehabil. 2015 Oct;94(10 Suppl 1):887-97. doi: 10.1097/PHM.0000000000000293. PMID 25888653